CLINICAL TRIAL: NCT00547183
Title: A Randomized, Double-Blind, Parallel-Design, Placebo-Controlled Study to Evaluate the Efficacy and Safety of Tadalafil (2.5 mg and 5 mg) Administered Once Daily to Men With Diabetes Mellitus and Erectile Dysfunction
Brief Title: Study the Safety and Effectiveness of Tadalafil in Men With Diabetes Who Have Problems Getting and Keeping an Erection
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: ICOS Corporation (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 8702; H6D-MC-LVFZ
Record Dates: First submitted 2007-10-18; First posted 2007-10-22 (Estimated); Last update posted 2007-10-22 (Estimated); Status verified 2007-10

CONDITIONS: Impotence
MeSH Terms: conditions — Erectile Dysfunction | interventions — Tadalafil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 2 (Active Comparator): 2.5 mg tadalafil
  Interventions: Drug: tadalafil
- 3 (Active Comparator): 5 mg tadalafil
  Interventions: Drug: tadalafil
- 1 (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: tadalafil — 2.5 mg tadalafil tablet taken by mouth once a day, no more than 1 dose a day, for 12 weeks
  Other Names: LY450190; Cialis; IC351
  Arms: 2
Drug: tadalafil — 5 mg tadalafil tablet taken by mouth once a day, no more than 1 dose a day, for 12 weeks
  Other Names: LY450190; Cialis; IC351
  Arms: 3
Drug: placebo — Placebo tablet taken by mouth once a day, no more than 1 dose per day, for 12 weeks
  Arms: 1

SUMMARY:
Study to evaluate the safety and effectiveness of 2.5 mg and 5 mg tadalafil when taken by men with diabetes mellitus who have problems getting and maintaining an erection.

ELIGIBILITY:
Inclusion Criteria:

* History of erectile dysfunction for at least 3 months.
* Currently have diabetes mellitus of at least 3 months duration.
* Agree to not use any other ED treatment during the study.
* Anticipate the same female sexual partner for the study.
* Must be willing to make the required number of sexual attempts.

Exclusion Criteria:

* History of other primary sexual disorder
* Treatment with nitrates or potent CYP3A4 inhibitors
* Have a penile implant or clinically significant penile deformity
* History of certain heart problems
* Have kidney or liver problems

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 298 (Actual)
Dates: Start 2004-10; Study Completion 2005-05 (Actual)

PRIMARY OUTCOMES:
Effectiveness measured by IIEF score of questions 1-5 and 15 plus the percentages of positive responses to questions 2 and 3 in the SEP diary | 12 weeks

SECONDARY OUTCOMES:
Change in the GAQ, SEP, IIEF, SEAR, and RSE scores. | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern Time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Genthin, Germany

REFERENCES:
- [Derived] Porst H, Gacci M, Buttner H, Henneges C, Boess F. Tadalafil once daily in men with erectile dysfunction: an integrated analysis of data obtained from 1913 patients from six randomized, double-blind, placebo-controlled, clinical studies. Eur Urol. 2014 Feb;65(2):455-64. doi: 10.1016/j.eururo.2013.09.037. Epub 2013 Oct 2. PMID 24119319
- [Derived] Shabsigh R, Seftel AD, Kim ED, Ni X, Burns PR. Efficacy and safety of once-daily tadalafil in men with erectile dysfunction who reported no successful intercourse attempts at baseline. J Sex Med. 2013 Mar;10(3):844-56. doi: 10.1111/j.1743-6109.2012.02898.x. Epub 2012 Oct 4. PMID 23035781
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com